CLINICAL TRIAL: NCT06183216
Title: A Randomized, Double Blinded, Positive Controlled Phase Ⅰb Clinical Trial in Participants Aged 2 Months (42-89 Days) and 2 to 5 Years to Evaluate the Safety and Immunogenicity of 13-valent Pneumococcal Polysaccharide Conjugate Vaccine
Brief Title: A Phase 1b Clinical Trial of 13-valent Pneumococcal Polysaccharide Conjugate Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sinovac Research and Development Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sinovac Biotech Co., Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PRO-PCV-1002
Record Dates: First submitted 2023-12-13; First posted 2023-12-27 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Pneumococcal Infectious Disease
MeSH Terms: conditions — Pneumococcal Infections | interventions — 13-valent pneumococcal vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Infants aged 2 months in experimental group (Experimental): 35 participants aged 2 months will be randomized to receive Sinovac PCV13. Route of administration is intramuscular injection at anterolateral aspect of thigh; immunization schedule is 4 doses, including 3 doses (two-month interval) in primary vaccination and a booster dose at the age of 12-15 months.
  Interventions: Biological: Sinovac PCV13
- Infants aged 2 months in control group (Active Comparator): 35 participants aged 2 months will be randomized to receive PREVNAR 13. Route of administration is intramuscular injection at anterolateral aspect of thigh; immunization schedule is 4 doses, including 3 doses (two-month interval) in primary vaccination and a booster dose at the age of 12-15 months.
  Interventions: Biological: PREVNAR 13
- Children aged 2-5 years in experimental group (Experimental): 35 children aged 2-5 years will be randomized to receive Sinovac PCV13. The route of administration is intramuscular injection at deltoid muscle of the upper arm, and immunization schedule is 1 dose for children aged 2-5 years old.
  Interventions: Biological: Sinovac PCV13
- Children aged 2-5 years in control group (Active Comparator): 35 children aged 2-5 years will be randomized to receive PREVNAR 13. The route of administration is intramuscular injection at deltoid muscle of the upper arm, and immunization schedule is 1 dose for children aged 2-5 years old.
  Interventions: Biological: PREVNAR 13

INTERVENTIONS:
Biological: Sinovac PCV13 — 0.5 mL dose of Sinovac PCV13 contains 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F saccharides.
  Arms: Children aged 2-5 years in experimental group; Infants aged 2 months in experimental group
Biological: PREVNAR 13 — 0.5 mL dose of PREVNAR 13 contains 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F saccharides.
  Arms: Children aged 2-5 years in control group; Infants aged 2 months in control group

SUMMARY:
A phase 1b clinical trial of 13-valent Pneumococcal Polysaccharide Conjugate Vaccine (PCV13) developed by Sinovac Life Science Co., Ltd will be conducted in children aged 2 months (42-89 days) and 2 to 5 years. The objective of the study is to evaluate the safety and immunogenicity of Sinovac PCV13. The trial is a randomized, double blinded, positive controlled study.

DETAILED DESCRIPTION:
A phase Ⅰb clinical trial of the study of 13-valent Pneumococcal Polysaccharide Conjugate Vaccine (PCV13) developed by Sinovac Life Science Co., Ltd (Sinovac) will be conducted in Chinese children aged 2 months (42-89 days) and 2 to 5 years. The trial is an randomized, double-blind and active controlled study. The objective of this study is to evaluate the safety and immunogenicity of PCV13 manufactured by Sinovac Life Science Co., Ltd. The active control vaccine is the PREVNAR 13 manufactured by Pfizer Inc. A total of 140 participants will be enrolled, including 70 children aged 2-5 years old, and 70 infants aged 2 months (42-89 days). Participants will be randomized to receive either Sinovac PCV13 or Pfizer PCV13 in a 1:1 ratio. Children aged 2-5 years old will receive 1 dose; Infants aged 2 months will receive 4 doses, including 3 doses (two-month interval) in primary vaccination and a booster dose at the age of 12-15 months.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy infants aged 2 months (42-89 days); Healthy children aged 2-5 years.
2. Proven vaccination certificate, birth certificate and legal identification documents
3. The participants' guardians can understand and voluntarily sign the informed consent form.
4. Participants and their guardians can obey requirements of the protocol.

Exclusion Criteria:

1. Received any pneumococcal vaccine prior to enrollment.
2. History of culture confirmed bacterial pneumonia or invasive pneumococcal disease (IPD) caused by Streptococcus pneumoniae.
3. History of allergy to the vaccine or vaccine components, including pneumococcal polysaccharide for each serotype, diphtheria CRM197, aluminum phosphate, succinic acid, polysorbate 80 and sodium chloride; or serious adverse reactions to the vaccine, such as urticaria, dyspnea, angioedema and asthma.
4. History of dystocia, asphyxia rescue, nervous system damage at birth (only applicable to infants aged 2 months (42-89 days))
5. Congenital malformations or developmental disorders, genetic defects, severe malnutrition, asthma etc.
6. Autoimmune disease (such as systemic lupus erythematosus) or immunodeficiency/ immunosuppression (such as HIV, organ transplantation)
7. Severe cardiovascular diseases, such as diabetes, liver diseases, kidney diseases, malignant tumors.
8. Family history of mental illness, severe neurological disease (epilepsy or convulsions) or mental illness.
9. History of thyroidectomy, asplenia, functional asplenia; and asplenia or splenectomy resulting from any condition.
10. Diagnosed abnormal blood coagulation function (eg, lack of blood coagulation factors, blood coagulopathy, abnormal platelets), history of obvious bleeding or bruising after intramuscular injection or venipuncture.
11. Infants 2 months of age (42-89 days) prior to enrollment/children 2 to 5 years of age 6 months prior to enrollment had been treated with corticosteroids, other immunosuppressive agents (excluding corticosteroid spray therapy for allergic rhinitis, superficial corticosteroid therapy for acute non-concurrent dermatitis) or cytotoxic therapy for ≥14 days
12. Infants 2 months of age (42-89 days) prior to enrollment/children 2 to 5 years of age 3 months prior to enrollment received blood products within the past 3 months (excluding hepatitis B immunoglobulin within 1 month).
13. Receipt of other investigational drugs in the past 60 days or have the plan to participate in other clinical trials during this study.
14. Receipt of attenuated live vaccines in the past 14 days.
15. Receipt of inactivated or subunit vaccines in the past 7 days.
16. Acute diseases or acute exacerbation of chronic diseases in the past 7 days.
17. Axillary temperature ≥37.3 °C.
18. According to the investigator's judgment, the subject has any other factors that are not suitable for participating in the clinical trial.

Ages: 6 Weeks to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 140 (Actual)
Dates: Start 2024-01-04 (Actual); Primary Completion 2025-03-26 (Actual); Study Completion 2025-03-26 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse reactions | 0-30 days after each dose
  Incidence of adverse reactions within 30 days after each dose

SECONDARY OUTCOMES:
Incidence of adverse reactions | 0-7 days after each dose
  Incidence of adverse reactions within 7 days after each dose
Incidence of SAE | 6 months after vaccination for children aged 2-5 years; 1 month after completion of booster vaccination for infants aged 2 months.
  Incidence of SAE during the period of safety monitoring
IgG concentration ≥0.35μg/mL for infants aged 2 months | 30 days after primary/booster immunization
  The proportion of participants achieving an IgG concentration ≥0.35μg/mL (seropositivity rate) for each serotype 30 days after primary/booster immunization.
IgG concentration ≥1.0μg/mL for infants aged 2 months | 30 days after primary/booster immunization
  The proportion of participants achieving an IgG concentration ≥1.0μg/mL for each serotype 30 days after primary/booster immunization.
GMCs for infants aged 2 months | 30 days after primary/booster immunization
  GMCs for each serotype 30 days after primary/booster immunization
GMIs for infants aged 2 months | 30 days after primary/booster immunization
  GMIs (GMC increase folds) for each serotype 30 days after primary/booster immunization
IgG concentration ≥0.35μg/mL for children aged 2-5 years | 30 days after vaccination
  The proportion of participants achieving an IgG concentration ≥0.35μg/mL (seropositivity rate) for each serotype 30 days after vaccination.
IgG concentration ≥1.0μg/mL for children aged 2-5 years | 30 days after vaccination
  The proportion of participants achieving an IgG concentration ≥1.0μg/mL for each serotype 30 days after vaccination.
GMCs for children aged 2-5 years | 30 days after vaccination
  GMCs for each serotype 30 days after vaccination
GMIs for children aged 2-5 years | 30 days after vaccination
  GMIs (GMC increase folds) for each serotype 30 days after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Yan Zheng, Principal Investigator — Yunnan Provincial Center for Disease Prevention and Control
Locations (1):
- Binchuan County Center for Diseases Control and Prevention, Dali, Yunnan, China